CLINICAL TRIAL: NCT04067336
Title: A Phase 1/2 First in Human Study of the Menin-MLL(KMT2A) Inhibitor KO-539 in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: First in Human Study of Ziftomenib in Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KO-MEN-001
Expanded Access: NCT05738538 (Available)
Record Dates: First submitted 2019-06-25; First posted 2019-08-26 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Advanced Malignant Neoplasm; Acute Myeloid Leukemia; Mixed Lineage Leukemia; Mixed Lineage Acute Leukemia; Acute Leukemia of Ambiguous Lineage; Mixed Phenotype Acute Leukemia; Acute Lymphoblastic Leukemia
Keywords: AML; Hematological malignancy; KMT2A; NPM1; Menin; Leukemia; Acute Leukemia; ALL; MLL; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; MEIS1
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hematologic Neoplasms; Leukemia | interventions — Midazolam; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1a - Dose Escalation (Experimental): AML patients will receive multiple doses of ziftomenib
  Interventions: Drug: Ziftomenib
- Phase 1b - Dose-Validation Expansion (Experimental): Cohort 1: KMT2A-r / NPM1-m R/R AML patients will receive ziftomenib
  Cohort 2: KMT2A-r / NPM1-m R/R AML patients will receive ziftomenib
  Interventions: Drug: Ziftomenib
- Phase 2 (Experimental): NPM1-m R/R AML patients will receive the recommended phase 2 ziftomenib dose
  Interventions: Drug: Ziftomenib
- Sub-study 1 (Experimental): R/R AML patients with mutations associated with MEIS1 overexpression will receive ziftomenib + midazolam
  Interventions: Drug: Ziftomenib; Drug: Midazolam
- Sub-study 2 (Experimental): R/R AML patients with mutations associated with MEIS1 overexpression will receive ziftomenib + itraconazole
  Interventions: Drug: Ziftomenib; Drug: Itraconazole
- Sub-study 3 (Experimental): Part 1a: KMT2A-r R/R ALL patients will receive multiple ziftomenib doses
  Part 1b: KMT2A-r R/R ALL patients will receive ziftomenib
  Interventions: Drug: Ziftomenib
- Sub-study 4 (Experimental): R/R AML patients with mutations associated with MEIS1 overexpression will receive ziftomenib
  Interventions: Drug: Ziftomenib

INTERVENTIONS:
Drug: Ziftomenib — Oral administration
  Other Names: KO-539
Drug: Midazolam — Oral administration
  Other Names: Seizalam; Hypnovel; Dormicum
  Arms: Sub-study 1
Drug: Itraconazole — Oral administration
  Other Names: Sporanox; Onmel; Tolsura
  Arms: Sub-study 2

SUMMARY:
In this trial, ziftomenib, a menin-MLL(KMT2A) inhibitor, will be tested in patients for the first time. The trial includes a Main Study and four sub-studies. In the Main Study (including Phase 1a, Phase 1b, and Phase 2 portions), ziftomenib will be evaluated in patients with relapsed or refractory (R/R) acute myeloid leukemia (AML). The main study has completed enrollment.

In Sub-studies 1 and 2, the effects of taking ziftomenib and other common drugs at the same time will be investigated in AML patients. In Sub-study 3, ziftomenib will be evaluated in patients with R/R acute lymphoblastic leukemia (ALL). In Sub-study 4, ziftomenib will be evaluated in patients with R/R AML with certain genetic mutations.

DETAILED DESCRIPTION:
This first-in-human (FIH), open-label study will assess ziftomenib, a menin-MLL(KMT2A) inhibitor, in patients with relapsed or refractory (R/R) acute myeloid leukemia (AML). The trial includes a Main Study and four sub-studies.

The Main Study is a Phase 1/2 dose-escalation and dose-validation/expansion study to assess ziftomenib in patients with R/R AML. The dose-escalation part of the study (Phase 1a) will determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D). The dose-validation/expansion part of the study (Phase 1b) will determine the safety, tolerability, and minimal biologically effective dose (MBED) of ziftomenib in biomarker-specific dosing cohorts from among doses that demonstrated early biological activity and are determined to be safe in the dose-escalation phase. The Phase 2 portion of the study will determine the safety, tolerability, and anti-leukemia activity of ziftomenib in patients with nucleophosmin 1-mutant (NPM1-m) AML.

In Sub-study 1, the effects of co-administration of ziftomenib on the pharmacokinetics (PK) of midazolam will be studied in patients with R/R AML with certain genetic mutations.

In Sub-study 2, the effects of co-administration of itraconazole on the PK of ziftomenib will be studied in patients with R/R AML with certain genetic mutations.

In Sub-study 3, the safety, tolerability, and MBED/RP2D of ziftomenib will be studied in patients with R/R KMT2A-rearranged (KMT2A-r) ALL (Phase 1a dose escalation). These parameters will be investigated further for the RP2D in a Phase 1b dose-validation/cohort expansion part of the sub-study.

In Sub-study 4, the clinical activity of ziftomenib will be studied in patients with R/R AML with certain genetic mutations.

ELIGIBILITY:
Key Inclusion Criteria:

Patients with refractory or relapsed AML defined as the reappearance of ≥ 5% blasts in the bone marrow and who have also failed or are ineligible for any approved standard of care therapies, including HSCT.

1. Phase 1b:

   * Patients with a documented lysine[K]-specific methyltransferase 2-rearrangement (KMT2A-r), or
   * Patients with a documented nucleophosmin 1 mutation (NPM1-m)
2. Phase 2:

   * Patients with a documented nucleophosmin 1 mutation (NPM1-m)
3. Sub-studies:

   * Sub-studies 1 and 2: Patients with R/R AML with NPM1-m or other mutations associated with MEIS1 overexpression.
   * Sub-study 3: Patients with R/R Acute Lymphoblastic Leukemia (ALL) with KMT2A-r.
   * Sub-study 4: Patients with R/R AML with mutations associated with MEIS1 overexpression.
4. ≥ 18 years of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2, and a life expectancy of at least 2 months.
6. Adequate liver and kidney function according to protocol requirements.
7. Peripheral white blood cell (WBC) counts ≤ 30,000/μL. Patients may receive hydroxyurea to control and maintain white blood cell count prior to enrollment.
8. Women of childbearing potential must be willing to use a highly effective method of contraception throughout the study and for at least 187 days after the last dose of study treatment.
9. Males with female partners of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least 97 days after the last dose of study treatment.

Key Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia.
2. Diagnosis of chronic myelogenous leukemia in blast crisis.
3. Donor lymphocyte infusion < 30 days prior to study entry.
4. Clinically active central nervous system (CNS) leukemia.
5. Undergone HSCT and have not had adequate hematologic recovery.
6. Receiving immunosuppressive therapy post HSCT within 2 weeks of Cycle 1 Day 1.
7. Grade ≥ 2 active graft-versus-host disease (GVHD), moderate or severe limited chronic GVHD, or extensive chronic GVHD of any severity.
8. Received chemotherapy immunotherapy, radiotherapy, or any ancillary therapy that is considered to be investigational (i.e., used for non-approved indications(s) and in the context of a research investigation) < 14 days prior to the first dose of ziftomenib or within 5 drug half-lives prior to the first dose of study drug.
9. Not recovered to < Grade 2 (National Cancer Institute Common Terminology Criteria for Adverse Events v5.0) from all acute toxicities or deemed back to a stable baseline.
10. Treatment with concomitant drugs that are strong inhibitors or inducers of cytochrome P450-isozyme 3A4 (CYP3A4), as follows:

    * Phase 1a, 1b, 2, and sub-studies 3 and 4: with the exception of antibiotics, antifungals, and antivirals that are used as standard of care or to prevent or treat infections and other such drugs that are considered absolutely essential for the care of the patient.
    * Sub-studies 1 and 2: No exceptions will be allowed except for the use of moderate CYP3A4 antifungal prophylaxis such as fluconazole or isavuconazole which is at steady state on Cycle 1 Day 1 and will continue through the completion of PKs on Cycle 1 Day 15 (for sub-study 1) or Cycle 1 Day 18 (for sub-study 2).
11. Detectable viral load for human immunodeficiency virus, hepatitis C, or hepatitis B surface antigen indicative of active infection. Patients with controlled disease will not be excluded from study enrollment.
12. Pre-existing disorder predisposing the patient to a serious or life-threatening infection (e.g. cystic fibrosis, congenital or acquired immunodeficiency, bleeding disorder, or cytopenias not related to AML).
13. Active uncontrolled acute or chronic systemic fungal, bacterial, viral, or other infection.
14. Significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension or arrhythmia, history of cerebrovascular accident including transient ischemic attack within the past 6 months, congestive heart failure (NYHA Class III or IV) related to primary cardiac disease, ischemic or severe valvular heart disease, or a myocardial infarction within 6 months prior to the first dose of study treatment.
15. Mean QTcF >480 ms on triplicate ECG.
16. Major surgery within 4 weeks prior to the first dose of study treatment.
17. Women who are pregnant or lactating. All female patients with reproductive potential must have a negative serum pregnancy test within 72 hours prior to starting treatment.
18. For sub-studies 1 and 2: Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of ziftomenib until the end of Cycle 1.
19. For sub-studies 1 and 2: Moderate (Child-Pugh class B) or severe (Child-Pugh class C) hepatic impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2028-10-16 (Estimated); Study Completion 2028-10-16 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) | Dose Limiting Toxicities (DLTs) will be evaluated during the first 28 days (1 cycle)
  MTD is defined as the highest dose that is not expected to cause dose limiting toxicity (DLT) in more than 20% of patients.
Phase 1b: Number of patients who experience Adverse Events (AEs) and Serious Adverse Events (SAEs) | During treatment and up to approximately 28 days after treatment discontinuation, or until immediately before the initiation of another anticancer therapy, whichever occurs first.
  Assessed by NCI-CTCAE v5.0
Phase 1b: Minimum biologically effective dose | For at least 12 months following end of treatment
  Minimum biologically effective dose in dosing cohorts which have demonstrated biological activity and have been determined to be safe as a part of Part 1a
Phase 1a, 1b, and 2: Evidence of anti-leukemia activity | For at least 12 months following end of treatment
  Assessed by the CR + CRh rate
Sub-study 1: Time to observed maximum plasma concentration (Tmax) of ziftomenib and midazolam | Cycle 1 on Days 1 and 15 at predose and postdose
  Tmax of ziftomenib, its metabolites, midazolam, and 1-hydroxymidazolam
Sub-study 1: Area under the plasma concentration-time curve from time 0 to time t (AUC0-t) of ziftomenib and midazolam | Cycle 1 on Days 1 and 15 at predose and postdose
  AUC0-t of ziftomenib, its metabolites, midazolam, and 1-hydroxymidazolam
Sub-study 1: Maximum observed plasma concentration (Cmax) of ziftomenib and midazolam | Cycle 1 on Days 1 and 15 at predose and postdose
  Cmax of ziftomenib, its metabolites, midazolam, and 1-hydroxymidazolam
Sub-study 2: Time to observed maximum plasma concentration (Tmax) of ziftomenib and itraconazole | Cycle 1 on Days 1, 15, and 22 at predose and postdose
  Tmax of ziftomenib, its metabolites, and itraconazole
Sub-study 2: Area under the plasma concentration-time curve from time 0 to time t (AUC0-t) of ziftomenib and itraconazole | Cycle 1 on Days 1, 15, and 22 at predose and postdose
  AUC0-t of ziftomenib, its metabolites, and itraconazole
Sub-study 2: Maximum observed plasma concentration (Cmax) of ziftomenib and itraconazole | Cycle 1 on Days 1, 15, and 22 at predose and postdose
  Cmax of ziftomenib, its metabolites, and itraconazole
Sub-study 3: Minimum biologically effective dose (MBED) and/or the recommended Phase 2 dose (RP2D) | During treatment and up to approximately 28 days after treatment discontinuation, or until immediately before the initiation of another anticancer therapy, whichever occurs first
  Assessed by the number of patients that experience Adverse Events (AEs) and Serious Adverse Events (SAEs) per NCI-CTCAE v5.0
Sub-study 3: Minimum biologically effective dose (MBED) and/or the recommended Phase 2 dose (RP2D) | For at least 12 months following end of treatment
  Assessed by CR
Sub-study 3: Change in Eastern Cooperative Oncology Group (ECOG) status | Timeframe: from Baseline to End of Treatment
  To assess the change in ECOG status
Sub-study 3: Time to observed maximum plasma concentration (Tmax) of ziftomenib | Postdose on Cycle 1 Day 1 and Cycle 2 Day 1. Predose at Cycle 2 onwards
  Tmax of ziftomenib
Sub-study 3: Area under the plasma concentration-time curve from time 0 to time t (AUC0-t) of ziftomenib | Postdose on Cycle 1 Day 1 and Cycle 2 Day 1. Predose at Cycle 2 onwards
  AUC0-t of ziftomenib
Sub-study 3: Maximum observed plasma concentration (Cmax) of ziftomenib | Postdose on Cycle 1 Day 1 and Cycle 2 Day 1. Predose at Cycle 2 onwards.
  Cmax of ziftomenib
Sub-study 4: Complete remission (CR) and complete remission with partial hematologic recovery (CRh) | For at least 12 months following end of treatment
  To assess the CR+CRh rate

SECONDARY OUTCOMES:
Phase 1a and 2: Number of patients that experience Adverse Events (AEs) and Serious Adverse Events (SAEs) | During treatment and up to approximately 28 days after treatment discontinuation, or until immediately before the initiation of another anticancer therapy, whichever occurs first.
  Assessed by NCI-CTCAE v5.0
Phase 1a: Tmax | Cycle 1 and Cycle 2. Each cycle is 28 days.
  Time to observed maximum plasma concentration of ziftomenib and/or its metabolites
Phase 1a: AUC(0-t) | Cycle 1 and Cycle 2. Each cycle is 28 days.
  Area under the plasma concentration-time curve from time 0 to time t of ziftomenib and/or its metabolites
Phase 1a: Cmax | Cycle 1 and Cycle 2. Each cycle is 28 days.
  Maximum plasma concentration of ziftomenib and/or its metabolites
Phases 1a, 1b, and 2: Complete remission (CR) and complete remission with partial hematologic recovery (CRh) measurable residual disease (MRD) negativity | For at least 12 months following discontinuation of treatment
  To assess the CR/CRh MRD negativity
Phases 1a, 1b, and 2: Duration of response (DOR) | For at least 12 months following discontinuation of treatment
  To assess the DOR, defined as the duration of CR/CRh
Phases 1a, 1b, and 2: Transfusion independence (TI) | For at least 12 months following discontinuation of treatment
  To assess transfusion independence
Phases 1a, 1b, and 2: Overall response rate (ORR) | For at least 12 months following discontinuation of treatment
  To assess the ORR
Phases 1a, 1b, and 2: Event-free survival (EFS) | For at least 12 months following end of treatment
  To assess event-free survival
Phases 1a, 1b, and 2: Overall survival (OS) | For at least 12 months following end of treatment
  To assess overall survival
Phases 1a, 1b, and 2: Composite complete remission (CRc) | For at least 12 months following discontinuation of treatment
  To assess CRc
Phases 1b and 2: Composite complete remission (CRc) measurable residual disease (MRD) negativity | For at least 12 months following discontinuation of treatment
  To assess the CRc MRD negativity
Phases 1b and 2: Overall response rate (ORR) measurable residual disease (MRD) negativity | For at least 12 months following discontinuation of treatment
  To assess the ORR MRD negativity
Sub-study 2: Corrected QT (QTc) intervals | During Cycle 1
  Assessed by QTc intervals
Sub-study 3: Complete remission (CR) measurable residual disease (MRD) negativity | For at least 12 months following discontinuation of treatment
  To assess the CR MRD negativity
Sub-studies 3 and 4: Composite complete remission (CRc) | For at least 12 months following discontinuation of treatment
  To assess CRc
Sub-study 3: Duration of response (DOR) | For at least 12 months following discontinuation of treatment
  To assess the DOR, defined as the duration of CR
Sub-studies 3 and 4: Overall survival (OS) | For at least 12 months following discontinuation of treatment
  To assess overall survival
Sub-studies 3 and 4: Event-free survival (EFS) | For at least 12 months following discontinuation of treatment
  To assess event-free survival
Sub-study 4: Transfusion independence (TI) | For at least 12 months following discontinuation of treatment
  To assess transfusion independence
Sub-studies 3 and 4: Overall response rate (ORR) measurable residual disease (MRD) negativity | For at least 12 months following discontinuation of treatment
  To assess the ORR MRD negativity
Sub-study 4: Number of patients that experience Adverse Events (AEs) and Serious Adverse Events (SAEs) | During treatment and up to approximately 28 days after treatment discontinuation, or until immediately before the initiation of another anticancer therapy, whichever occurs first.
  Assessed by NCI-CTCAE v5.0
Sub-study 4: Duration of response (DOR) | For at least 12 months following discontinuation of treatment
  To assess the DOR, defined as the duration of CR/CRh
Sub-study 4: Time to observed maximum plasma concentration (Tmax) of ziftomenib | Postdose on Cycle 1 Day 1 and Cycle 2 Day 1. Predose on Cycle 2 onwards
  Tmax of ziftomenib and its metabolites
Sub-study 4: Area under the plasma concentration-time curve from time 0 to time t (AUC0-t) of ziftomenib | Postdose on Cycle 1 Day 1 and Cycle 2 Day 1. Predose on Cycle 2 onwards
  AUC0-t of ziftomenib and its metabolites
Sub-study 4: Maximum plasma concentration (Cmax) of ziftomenib | Postdose on Cycle 1 Day 1 and Cycle 2 Day 1. Predose on Cycle 2 onwards
  Cmax of ziftomenib and its metabolites

CONTACTS AND LOCATIONS:
Locations (56):
- United States (23):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack University Medical Center - John Theurer Cancer Center, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Weill Cornell Medical College - NY Presbyterian Hospital, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Oklahoma University Health - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Harold C. Simmons Comprehensive Cancer Center - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Belgium (3):
  - UZ Brussel, Jette
  - AZ Delta - Campus Rumbeke, Roeselare
  - CHU UCL Namur, Yvoir
- Canada (4):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - McMaster University Juravinski Cancer Centre, Hamilton, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Hopital de l'Enfant-Jesus - Centre Integre en Cancerologie du CHU de Quebec - Universite Laval, Québec, Quebec
- France (6):
  - Centre Hospitalier Universitaire de Lille, Lille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Hopital Saint Louis, Paris
  - Magendie Hopital Haut-Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Charitè-Campus Benjamin Franklin, Berlin
  - University Medicine Greifswald, Greifswald
  - Medizinische Hochsschule Hannover, Hanover
  - Johannes Gutenberg - University Mainz, Mainz
- Italy (4):
  - Institute of Hematology and Medical Oncology "L. and A. Seragnoli", Bologna
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori", Meldola
  - UO Ematologia Ospedale di Ravenna, Ravenna
  - Institution Fondazione Policlinico Tor Vergata, Roma
- Nasz Lekarz Przychodnie Medyczne, Torun, Poland
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Universitat de Barcelona, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (4):
  - Cardiff and Vale University, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Barts Health NHS Trust, London
  - St. George's Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang ES, Montesinos P, Foran J, Erba H, Rodriguez-Arboli E, Fedorov K, Heiblig M, Heidel FH, Altman JK, Baer MR, Ades L, Pettit K, Peterlin P, Papayannidis C, Berthon C, Walter RB, Shah MV, Balasubramanian S, Khawandanah M, Salamero Garcia O, Bergeron J, Madanat YF, Roboz GJ, Ulrickson M, Redner RL, McCloskey J, Pigneux A, de la Fuente Burguera A, Mitra A, Soifer HS, Tabachri M, Zhang Z, Riches M, Corum D, Leoni M, Issa GC, Fathi AT; KOMET-001. Ziftomenib in Relapsed or Refractory NPM1-Mutated AML. J Clin Oncol. 2025 Nov;43(31):3381-3390. doi: 10.1200/JCO-25-01694. Epub 2025 Sep 25. PMID 40997296
- [Derived] Wang ES, Issa GC, Erba HP, Altman JK, Montesinos P, DeBotton S, Walter RB, Pettit K, Savona MR, Shah MV, Kremyanskaya M, Baer MR, Foran JM, Schiller G, Ades L, Heiblig M, Berthon C, Peterlin P, Rodriguez-Arboli E, Salamero O, Patnaik MM, Papayannidis C, Grembecka J, Cierpicki T, Clegg B, Ray J, Linhares BM, Nie K, Mitra A, Ahsan JM, Tabachri M, Soifer HS, Corum D, Leoni M, Dale S, Fathi AT. Ziftomenib in relapsed or refractory acute myeloid leukaemia (KOMET-001): a multicentre, open-label, multi-cohort, phase 1 trial. Lancet Oncol. 2024 Oct;25(10):1310-1324. doi: 10.1016/S1470-2045(24)00386-3. PMID 39362248
- [Derived] Sasca D, Guezguez B, Kuhn MWM. Next generation epigenetic modulators to target myeloid neoplasms. Curr Opin Hematol. 2021 Sep 1;28(5):356-363. doi: 10.1097/MOH.0000000000000673. PMID 34267079
- [Derived] Jimenez JA, Apfelbaum AA, Hawkins AG, Svoboda LK, Kumar A, Ruiz RO, Garcia AX, Haarer E, Nwosu ZC, Bradin J, Purohit T, Chen D, Cierpicki T, Grembecka J, Lyssiotis CA, Lawlor ER. EWS-FLI1 and Menin Converge to Regulate ATF4 Activity in Ewing Sarcoma. Mol Cancer Res. 2021 Jul;19(7):1182-1195. doi: 10.1158/1541-7786.MCR-20-0679. Epub 2021 Mar 19. PMID 33741715